CLINICAL TRIAL: NCT03801226
Title: Zero Sodium Peritoneal Dialysate Protocol in Human Pilot Study
Brief Title: Zero Sodium Peritoneal Dialysate Protocol Pilot Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Jeffrey Testani, Associate Professor of Medicine, Yale University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2000023570
Record Dates: First submitted 2018-12-12; First posted 2019-01-11 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Potential Applications for Heart Failure; Volume Overload
Keywords: Peritoneal dialysis
MeSH Terms: conditions — Edema | interventions — Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 10% dextrose in sterile water (Experimental): Patients randomized to this arm will undergo a two-hour dwell with 10% dextrose in sterile water at their first visit and Dianeal Low-Calcium with 4.25% Dextrose at their second visit.
  Interventions: Drug: Two-hour dwell with 10% dextrose in sterile water; Drug: Two-hour dwell with Dianeal Low-Calcium with 4.25% Dextrose
- Dianeal Low-Calcium with 4.25% Dextrose (Active Comparator): Patients randomized to this arm will undergo a two-hour dwell with Dianeal Low-Calcium with 4.25% Dextrose at their first visit and 10% dextrose in sterile water at their second visit.
  Interventions: Drug: Two-hour dwell with 10% dextrose in sterile water; Drug: Two-hour dwell with Dianeal Low-Calcium with 4.25% Dextrose

INTERVENTIONS:
Drug: Two-hour dwell with 10% dextrose in sterile water — Patients will be randomized to undergo a two-hour dwell with 10% dextrose in sterile water at their first or second study visit and will receive the alternate intervention at the other study visit.
Drug: Two-hour dwell with Dianeal Low-Calcium with 4.25% Dextrose — Patients will be randomized to undergo a two-hour dwell with Dianeal Low-Calcium with 4.25% Dextrose at their first or second study visit and will receive the alternate intervention at the other study visit.

SUMMARY:
The following pilot study will be undertaken to determine the effects of use of a zero-sodium peritoneal dialysate solution (10% dextrose in sterile water) on sodium removal as compared to a standard peritoneal dialysis solution.

DETAILED DESCRIPTION:
While heart failure (HF) is generally regarded as the inability of the heart to pump sufficient blood, on a population level, volume overload is the primary driver of morbidity and hospitalization. The signs and symptoms of volume overload are driven by water accumulation, which is initially driven by sodium retention. This overall goal of this study is to investigate the ability to remove sodium through use of a zero-sodium solution in peritoneal dialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients actively undergoing peritoneal dialysis (PD) with a functioning PD catheter
2. PD vintage < 3 years
3. As judged by treating nephrologist to be at or above optimal volume status (i.e., not dehydrated)

Exclusion Criteria:

1. Uncontrolled diabetes with frequent episodes of severe hyperglycemia
2. Systolic blood pressure < 100 mmHg
3. Serum sodium < 130 mEq/L
4. 1 or more episodes of peritonitis in the previous 6 months or active infection of the peritoneal dialysis catheter
5. Anemia with hemoglobin <8 g/dL
6. Serum bicarbinate < 18 mEq/L
7. Anuric renal failure
8. Inability to give written informed consent or follow study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability measured by protocol discontinuation due to patient discomfort or adverse event | Two hours
  Protocol discontinuation will be defined by premature draining of the 10% dextrose peritoneal solution (or 4.25% standard PD solution) prior to the planned two hour drain.

SECONDARY OUTCOMES:
Comparison of total sodium removed compared to baseline | Two hours
  This exploratory efficacy outcome will be addressed by comparing the quantity of sodium removed during the two-hour dwell between the two solutions

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Rao VS, Turner JM, Griffin M, Mahoney D, Asher J, Jeon S, Yoo PS, Boutagy N, Feher A, Sinusas A, Wilson FP, Finkelstein F, Testani JM. First-in-Human Experience With Peritoneal Direct Sodium Removal Using a Zero-Sodium Solution: A New Candidate Therapy for Volume Overload. Circulation. 2020 Mar 31;141(13):1043-1053. doi: 10.1161/CIRCULATIONAHA.119.043062. Epub 2020 Jan 8. PMID 31910658